CLINICAL TRIAL: NCT04343859
Title: A Phase I Clinical Trial of IMMH-010 in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of IMMH-010 in Patients With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tianjin Chasesun Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-IMMH001
Record Dates: First submitted 2020-03-23; First posted 2020-04-13 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2022-12

CONDITIONS: Malignant Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMMH-010 (Experimental): After Dose escalation study, Dose expansion study will be conducted :
  360mg and above,IMMH-010, QD or BID,Cycle1Day1-CycleN.
  Interventions: Drug: IMMH-010

INTERVENTIONS:
Drug: IMMH-010 — After tolerance study, 360mg and above IMMH-010 will be administered in Dose expansion study.

SUMMARY:
Phase I study of IMMH-010 in patients with advanced malignant solid tumors

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of single-dose and multi-dose IMMH-010 in patients with advanced solid tumors, et al.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible only if they meet all the following criteria:

1. Age ≥ 18 years when they sign the informed consent form;
2. Patients with advanced or metastatic solid tumors that are confirmed by cytological or histological examination, who did not respond to standard treatment regimens, or did not tolerate these regimens, or had no effective standard treatment regimens, or refused standard treatment regimens;
3. The ECOG score is 0 or 1 point (see the scoring criteria in Appendix 1);
4. Based on RECIST 1.1 (see the scoring criteria in Appendix 4), Subjects in Part B study must have at least one measurable lesion, and subjects in Part A study may have no measurable lesion;

   Definition of measurable lesion:
   1. Tumor lesion: The size must be accurately measurable on two mutually perpendicular diameters, and both diameters must be ≥10 mm or ≥2 times of the slice thickness
   2. Lymph node lesion: The size must be accurately measurable on two mutually perpendicular diameters, and both diameters must be ≥15 mm or ≥2 times of the slice thickness
5. In subjects who had received other treatments, the toxic and side effects should return to grade ≤ 1 or to the baseline (NCI-CTCAE 5.0, excluding alopecia);
6. The expected survival time should be at least 3 months;
7. Subjects should have appropriate organ and bone marrow functions, and have laboratory test results within the following ranges before entering the group:

   Bone marrow reserve (within 14 days, no transfusion of blood or blood products, or no correction by G-CSF or other hematopoietic stimulate factors): absolute neutrophils count (ANC) ≥1.5×109/L; hemoglobin (HB) ≥90 g/L; and platelet (PLT) ≥75×109/L; Liver function: ALT≤2.5×ULN; AST≤2.5×ULN; ALP≤2.5×ULN; TBIL≤1.5×ULN (patients with known Gilbert's disease are eligible if their serum bilirubin level ≤3×ULN; and patients with metastases to liver are eligible if their ALT≤5×ULN, AST≤5×ULN, and ALP≤5×ULN); and albumin ≥3 g/dL; Kidney function: creatinine ≤1.5×ULN or creatinine clearance ≥45 mL/min as calculated according to Cockcroft-Gault formula (refer to Appendix 2); Blood coagulation function: INR, PT, and APTT≤1.5×ULN (in patients not on anticoagulants; and it is decided by investigators whether patients on anticoagulants are eligible); Cardiac enzymes CK and CKMB measures are not exceeding the upper limit of normal value; Thyroid function measures are within the normal range or mildly abnormal but requiring no treatment.
8. Fertile eligible patients (males and females) must give their consent to taking reliable contraceptive measures (hormone, barrier, or sexual abstinence) throughout the trial and at least 4 months after the last dosing; reproductive-age females must have negative blood or urine pregnancy test within 21 days prior to initial dosing;
9. The subjects must give their informed consent for the study and signed ICF voluntarily before the trial;
10. The subjects or the statutory agents should be able to communicate well and complete the study complying with the protocol.

Exclusion Criteria:

Subjects are excluded if they meet one of the following exclusion criteria.

1. Subjects with a past history of pulmonary fibrosis or interstitial pneumonia, including pneumoconiosis or radiation fibrosis of lung beyond the exposure field, which is clinically significant as judged by the investigators;
2. Subjects who have received systemic glucocorticoid or any immunosuppressive agents for some condition within 14 days prior to the initial dosing, excluding local glucocorticoid via nose spray, aspiration, or other route, or systemic glucocorticoid at a physiological dose (namely not exceeding 10 mg/d of prednisone or an equivalent dose of other glucocorticoids); corticosteroids are allowed in subjects for pretreatment for venous contrast agent allergic reaction (scanning-relevant) in the study period, but it should be recorded.
3. Subjects who are expected to receive other systemic antineoplastic treatments in the study period;
4. Subjects with risks of intestinal obstruction or intestinal perforation, such as a history of diverticulitis, intra-abdominal abscess, active ulcer, GI tract obstruction, or abdominal cancer;
5. Subjects who are diagnosed with other malignant tumors within 5 years prior to the initial dosing, excluding eradicated basal cell carcinoma of skin, squamous cell carcinoma of skin, and / or radically resected in situ cancer;
6. Subjects who ever received any organ transplants, including allogeneic stem cell transplantation, but excluding those requiring no immunosuppression (such as corneal transplant and hair transplant);
7. Subjects with active metastasis to CNS and / or carcinomatous meningitis (including leptomeningeal carcinomatosis) with clinical symptoms or requiring intervention, which is unsuitable for the subjects to enter the group as judged by the investigators;
8. Subjects with active autoimmune diseases in the past 1 year and consequently requiring systemic treatments (namely systemic steroids or immunosuppressive agents);
9. Dysphagia affects oral dosing;
10. Subjects with refractory third lacunar effusion, such as massive pleural effusion and ascites;
11. Subjects with gastrointestinal disorders that might affect drug absorption (such as Crohn's disease, ulcerative colitis, and subtotal gastrectomy);
12. Subjects who received any immune checkpoint blockade therapy within 4 weeks or 5 drug half-lives (the shorter duration shall prevail), or the following immune-related adverse events (irAE) have occurred during the course of previous immunotherapy:

    a) Grade ≥3 immune-associated pneumonia; b) Grade ≥2 immune-related myocarditis;
13. Subjects who received major surgery within 4 weeks prior to the initial dosing or those whose wound did not completely heal yet; or subjects who received >30 Gy of chest radiotherapy within 6 months prior to the initial dosing;
14. Subjects with a history of myocarditis, myocardial infarction, cerebrovascular accident, or NHYA≥2 congestive cardiac failure within 6 months prior to the initial dosing; or subjects with uncontrollable angina, unstable angina, or uncontrollable arrhythmia;
15. Subjects who received other investigational drugs within 14 days or 5 half-lives (the longer duration shall prevail) prior to the initial dosing;
16. Subjects who were vaccinated with live vaccines within 30 days prior to the initial dosing, and live-virus-free influenza vaccines are allowed;
17. Subjects with active infections requiring systemic treatments (antibiotics); or subjects who meet any one of the following criteria:

    1. Subjects positive for human immunodeficiency virus (HIV) or with a known history of acquired immune deficiency syndrome
    2. Subjects with infection of hepatitis B virus (HBV) or hepatitis C virus (HCV) (definition: HBsAg-positive and HBV DNA copy number exceeding ULN, or HCV-Ab-positive);
    3. Subjects with active tuberculosis (with an exposure history or positive tuberculosis test, and with clinical and / or imaging manifestations).
    4. Subjects positive for treponema pallidum antibody.
18. Subjects with a history of serious hypersensitivity reaction of drug;
19. Pregnant or breast-feeding women;
20. Subjects who were ineligible to participate in clinical trials as judged by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Part A Dose escalation study at the end of Cycle 1 (Cycle1 is 21 days)
  To identify the dose-limiting toxicity (DLT) in dose escalation study.
Adverse reaction rate | From date of singing informed consent until the 30 days after the last study dose or the start date of a new anti-cancer therapy, whichever came first.
  Observe all the participants in any adverse events occurred during the period of clinical research, including clinical symptoms and signs of life, an abnormal in laboratory tests, record its clinical characteristics, severity, occurrence time, duration, treatment and prognosis, and determine its and the correlation between test drugs. NCI-CTCAE 5.0 standard was used to evaluate drug safety.

SECONDARY OUTCOMES:
Cmax | Part A Dose escalation study: At the end of Cycle1(Cycle1 is 21 days), Part B: At the end of Cycle0(Cycle0 is 4 days).
  Peak plasma concentration.
Tmax | Part A Dose escalation study: At the end of Cycle1(Cycle1 is 21 days), Part B: At the end of Cycle0(Cycle0 is 4 days).
  Time to peak plasma concentration.
AUC | Part A Dose escalation study: At the end of Cycle1(Cycle1 is 21 days), Part B: At the end of Cycle0(Cycle0 is 4 days).
  Area under the plasma concentration versus time curve.
Objective response rate (ORR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first (up to approximately 2 years).
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1.
Duration of response (DOR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first (up to approximately 2 years).
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression or death (whichever occurs first) as assessed by RECIST 1.1.
Disease control rate (DCR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first (up to approximately 2 years).
  DCR is defined as the percentage of participants who have BOR of CR or PR or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1.
Progression-free survival (PFS) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first (up to approximately 2 years).
  PFS is defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang J, Zou X, Liu Y, Liu X, Dong K, Yao X, Feng Z, Chen X, Sheng L, Li Y. Simultaneous Determination of a Novel PD-L1 Inhibitor, IMMH-010, and Its Active Metabolite, YPD-29B, in Rat Biological Matrices by Polarity-Switching Liquid Chromatography-Tandem Mass Spectrometry: Application to ADME Studies. Front Pharmacol. 2021 Jun 21;12:677120. doi: 10.3389/fphar.2021.677120. eCollection 2021. PMID 34234673